CLINICAL TRIAL: NCT01590563
Title: A Study to Evaluate the Safety and Initial Efficacy of a Spherical Copper Intrauterine Contraceptive Device the IUB(tm)
Brief Title: A Study to Evaluate the Safety and Initial Efficacy of a Novel Intrauterine Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocon Medical Ltd. (Industry)
Responsible Party: Principal Investigator, Dana Raveh Arbel, VP Clinical, Ocon Medical Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AOS-C1000-02
Record Dates: First submitted 2012-04-20; First posted 2012-05-03 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: Intrauterine device
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCu300A IUB (Experimental): Insertion of a spherical IUD (intrauterine device) with one year follow-up
  Interventions: Device: IUD

INTERVENTIONS:
Device: IUD — Insertion of a spherical IUD, one year follow-up
  Other Names: SCu300A IUB(tm)

SUMMARY:
Current intrauterine devices (IUD) pose such risks as uterine perforation during insertion, malposition and expulsion. The investigated device, the IUB(tm) SCu300A is an IUD which is inserted in a similar fashion into the uterus and takes a three dimensional spherical shape while curving away from the fundus. Apart for an anticipated reduction in the rate of stated complications, its smaller size and mallable characteristics are also expected to improve user experience. The clinical trial is intended to evaluate the safety and initial efficacy of this novel device.

DETAILED DESCRIPTION:
A copper IUD (intrauterine device or coil) is a type of intrauterine contraceptive device. Most IUDs have a plastic T-shaped frame which is wrapped in copper wire and sleeves. The device has to be fitted inside and removed from the uterine cavity by a doctor or qualified medical practitioner. It remains in place the entire time pregnancy is not desired.

The IUD is a long acting reversible contraceptive, with different IUDs intended to last for different lengths of time, usually between 3 and 10 years. The length of time that the device lasts depends mainly on the amount of exposed copper, which is indicated, in square millimeters, by a number in the name of each device (i.e., the Paragard T-380A has 380 square millimeters of exposed copper).

The IUD is the world's most widely used method of reversible birth control, currently used by over 175 million women.

The mechanism of IUDs is not well understood. It is known however that the presence of a device in the uterus prompts the release of leukocytes and prostaglandins by the endometrium. These substances are hostile to both sperm and eggs; the presence of copper increases the spermicidal effect. The general medical consensus is that spermicidal and ovicidal mechanisms are the only way in which IUDs work. Some physicians and medical texts have suggested they may have a secondary effect of interfering with the development of pre-implanted embryos; this secondary effect is considered more plausible when the IUD is used as emergency contraception.

Second-generation copper-T IUDs have failure rates of less than 1% per year, and cumulative 10-year failure rates of 2-6%. A copper IUD may also be used as emergency contraception. If an IUD is inserted within five days of unprotected intercourse, a woman's chance of pregnancy is reduced to that of ongoing IUD users.

IUDs do not protect against STDs or PID.

Made from a shape memory alloy of a specific size and shape, the SCu300A IUB™ is inserted through an insertion tube much like regular IUDs, however, when pushed out, in the uterus, it takes a spherical shape. An important feature includes its downwards curving opposite to the uterine fundus as it emerges out of the tube, minimizing the risk of perforation. The three dimensional shape's elasticity allows for better amenability to the uterus, nullifying the possibility of malposition and its final outer diameter reducing the probability of expulsion. Lacking rigid or protruding segments and being significantly smaller than other IUDs, the IUB™ is expected to reduce distortion and tissue irritation, possibly resulting in less bleeding, discomfort and pain, leading to lower discontinuation rates. A thread is attached to the IUB™ to allow easy removal.

The trialed IUB™ will be copper-based (Cu surface area of 300mm2).

This study aims to assess the IUB™'s safety and initial efficacy. Endpoints include the assessment of changes in discomfort, pain and menorrhea, changes in the endometrium discontinuation rates as well as user experience. These results will be used as regulatory evidence and will also help in reaffirming the assumption that the IUB™'s design contributes to lower complication and side effect rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult female aged 25-42
* Free willing to fully comply with treatment process
* Healthy women
* Married or in a steady relationship. Blood hemoglobin >11.5gr%
* Signed informed consent form

Exclusion Criteria:

* Pregnancy or suspicion of pregnancy
* Use of other contraception methods
* Abnormalities of the uterus resulting in distortion of the uterine cavity
* Acute current or past history of pelvic inflammatory disease, or current behavior suggesting a high risk for pelvic inflammatory disease
* Postpartum endometritis or postabortal endometritis in the past 3 months
* Known or suspected uterine or cervical malignancy
* Genital bleeding of unknown etiology
* Mucopurulent cervicitis
* Wilson's disease
* Allergy to any component of IUB™
* A previously placed IUD that has not been removed
* Known intolerance or allergy to copper and/or copper IUDs
* Medication that may interfere with the subject's ability to complete the protocol
* Any other significant disease or condition that could interfere with the subject's ability to complete the protocol
* A history of alcohol or drug abuse
* known infection with human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Planned pregnancy during the follow-up period
* Participation in another clinical trial
* Anemia of any kind or blood hemoglobin lower than 11.5gr%.

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beata Szoczei, MD, Principal Investigator — Synexus Hungary Kft.
Locations (1):
- Synexus Hungary Limited, Budapest, Hungary

REFERENCES:
- [Derived] Baram I, Weinstein A, Trussell J. The IUB, a newly invented IUD: a brief report. Contraception. 2014 Feb;89(2):139-41. doi: 10.1016/j.contraception.2013.10.017. Epub 2013 Nov 7. PMID 24309220

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCu300A IUB
Started | 15
Completed | 14
Not Completed | 1
Not completed — simple uterine hyperplasia - not related | 1

BASELINE CHARACTERISTICS:
Arm/Group | SCu300A IUB
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (4.8)
Sex/Gender, Customized [Number; unit: participants] | 15
Region of Enrollment [Number; unit: participants]
  Hungary | 15
Prior Contraception Use [Number; unit: participants]
  Yes | 8
  No | 7

OUTCOME MEASURES:

1. Primary Outcome: Rates of Uterine Perforation
Description: Uterine perforation is an established risk of IUD deployment which may cause certain health hazards. It is anticipated that the IUB(tm), through its form and deployment pattern, will reduce this risk.
Time Frame: During installation
Measure: Number; unit: Number of cases
Groups:
- Investigated Device Group: Group inserted the investigated device - the IUB SCu300A
Arm/Group | Investigated Device Group
Number analyzed (Participants) | 15
Number of cases | 0 [NR to 18.1%]

2. Primary Outcome: Efficacy in Preventing Pregnancy
Description: Prevention of pregnancy will be measured. Pregnancy rates are expected to be comparable to current IUDs.
Time Frame: 12 months
Measure: Number; unit: Number of pregnancies
Arm/Group | SCu300A IUB
Number analyzed (Participants) | 15
Number of pregnancies | 0

3. Secondary Outcome: Occurrence of Malposition, Expulsion.
Description: Expulsion and malposition are established risks involved with IUD use. Occurrence of these risks may drastically reduce effectiveness. It is expected that the IUB(tm) form will reduce these risks.
Time Frame: 12 months
Measure: Number; unit: Number of cases
Arm/Group | SCu300A IUB
Number analyzed (Participants) | 15
Number of cases | 0

ADVERSE EVENTS:
Arm/Group | SCu300A IUB
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCu300A IUB (N=15)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) — Investigated device was removed, condition not caused by investigated device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No